CLINICAL TRIAL: NCT07201428
Title: The Effects of Fiber Content in Enteral Nutrition Products on Opioid-Induced Constipation in Intubated Patients
Brief Title: Fiber-Enriched Enteral Nutrition and Opioid-Induced Constipation in the ICU
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Olcay Dilken, principal investigator, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: olcay-31
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Constipation, Opioid-Induced
Keywords: constipation; opioid; mechanical ventilation; sedation
MeSH Terms: conditions — Opioid-Induced Constipation; Constipation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Opioid use for sedation and analgesia is widespread among mechanically ventilated ICU patients, often leading to gastrointestinal dysfunction and opioid-induced constipation (OIC). While enteral nutrition (EN) is routinely used in critical care, the role of fiber-enriched EN formulas in preventing OIC remains unclear. This prospective quasi-randomized study aims to evaluate whether fiber-containing EN products reduce the incidence and severity of OIC compared to fiber-free formulations in intubated ICU patients. The findings may contribute to optimizing nutritional strategies to mitigate constipation-related complications in this high-risk population.

DETAILED DESCRIPTION:
The use of opioids for sedation and analgesia is common among intensive care unit (ICU) patients requiring mechanical ventilation. However, frequent and sometimes high-dose opioid administration can lead to gastrointestinal dysfunction and complications such as constipation. These complications are associated with increased risk of gastric content aspiration, suboptimal nutritional intake, prolonged ICU stays, and higher mortality rates.

Enteral nutrition (EN) is routinely administered to ICU patients unless there is a contraindication to gastrointestinal feeding . EN products are formulated with diverse compositions to address the needs of ICU patients, who represent a highly heterogeneous population. High-fiber EN formulations are typically used in patients with diarrhea or constipation. However, current literature lacks evidence regarding the efficacy of fiber-enriched EN in reducing constipation among intubated ICU patients.

In the study, the investigator aim to investigate whether high-fiber EN products have an effect on opioid-induced constipation compared to fiber-free products in intubated patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients over the age of 18 who are initiated on enteral nutrition and are on mechanical ventilation will be included in the study.

Exclusion Criteria:

* Pediatric and pregnant patients
* Life expectancy less than 24 hours
* Gastrointestinal surgery within the last week
* Intra-abdominal pressure > 15 mmHg
* Shock requiring high vasopressor support
* Contraindication to enteral nutrition
* Intubation >48 hours

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients over the age of 18 who are initiated on enteral nutrition and are on mechanical ventilation will be included in the study
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
the day of first defecation | 1-7 days
  The definition of first defecation was defined as stool volume >100 ml

SECONDARY OUTCOMES:
Need for enema use | 1-7 days
  Indication for constipation and need for enema use

CONTACTS AND LOCATIONS:
Locations (1):
- Sisli Hamidiye Etfal Training Hospital, Istanbul, Turkey (Türkiye)